CLINICAL TRIAL: NCT03641534
Title: Perfusion and Lung Congestion Evaluation Related to Fluids and Vasopressors in Sepsis and Malaria. (PERFuSE): an Observational Study
Brief Title: Monitoring of Perfusion in Sepsis and Malaria
Acronym: PERFuSE
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); University of Amsterdam (Other); University of British Columbia (Other); Chittagong Medical College and Hospital (Other); Malaria Research Group & Dev Care Foundation, Dhaka, Bangladesh (Unknown); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MAL18001
Record Dates: First submitted 2018-05-29; First posted 2018-08-22 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2020-09

CONDITIONS: Severe Sepsis; Malaria
Keywords: Perfusion; Lung congestion
MeSH Terms: conditions — Sepsis; Malaria | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hematocrit and peripheral blood parasitemia in thin and thick films will be assessed at T=0 (enrolment) then 6-hourly until parasite clearance (two consecutive negative thick smears per 500 white blood cells). Plasma creatinine will be measured 24-hourly for 72 hours, at discharge and day 14. Venous blood gas and lactate will be assessed 6-hourly until lactate <2 mmol/L.
  Arterial blood gas will be collected at T0 and after 24 hours if the subject is in respiratory distress, defined as respiratory rate > 30 breaths per minute and SpO2 <92% on room air. More frequent hematological and biochemical measurements may be done if clinically indicated at the discretion of the treating clinician. Plasma cell-free hemoglobin (CFH) will be analyzed at hour 0, 6, 24, 48, 72 and day 7 in the severe malaria group and only hour 0 in sepsis and uncomplicated malaria groups. Blood cultures and additional microbiology assays will be drawn at enrolment and performed locally.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sepsis
  Interventions: Procedure: Lung Ultrasound examination; Procedure: Compression ultrasonography (CUS); Procedure: Echocardiography; Procedure: Inferior Vena Cava ultrasound; Procedure: Passive leg raising test (PLR); Procedure: Orthogonal polarization spectral imaging (OPS); Procedure: Urine collection (Foley catheter); Procedure: Venous blood samplings; Procedure: Electrocardiogram; Procedure: GlycoCheck
- Severe malaria
  Interventions: Procedure: Lung Ultrasound examination; Procedure: Compression ultrasonography (CUS); Procedure: Echocardiography; Procedure: Inferior Vena Cava ultrasound; Procedure: Passive leg raising test (PLR); Procedure: Orthogonal polarization spectral imaging (OPS); Procedure: Urine collection (Foley catheter); Procedure: Venous blood samplings; Procedure: Electrocardiogram; Procedure: GlycoCheck
- Uncomplicated malaria
  Interventions: Procedure: Lung Ultrasound examination; Procedure: Compression ultrasonography (CUS); Procedure: Echocardiography; Procedure: Inferior Vena Cava ultrasound; Procedure: Passive leg raising test (PLR); Procedure: Orthogonal polarization spectral imaging (OPS); Procedure: Urine collection (Foley catheter); Procedure: Venous blood samplings; Procedure: Electrocardiogram; Procedure: GlycoCheck

INTERVENTIONS:
Procedure: Lung Ultrasound examination — Use of lung ultrasound to detect pulmonary complications
Procedure: Compression ultrasonography (CUS) — CUS is a highly sensitive and specific modality used to recognize lower extremity deep venous thrombosis (DVT)
Procedure: Echocardiography — Echocardiogram can be (i) identify imminent life-threatening causes of hemodynamic failure, (ii) recognize coexisting diagnoses that complicate management, (iii) follow the evolution of the disease process, and (iv) monitor response to treatment
Procedure: Inferior Vena Cava ultrasound — Measurement of the inferior vena cava diameter
Procedure: Passive leg raising test (PLR) — Baseline assessment (including pulse rate, systolic and diastolic blood pressure, velocity time integral (VTI) and stroke volume (SV) echocardiographic measurements) will be performed in the resting semi-recumbent position, defined as a position with the trunk elevated 30° to 45° relative to the lower limbs.
Procedure: Orthogonal polarization spectral imaging (OPS) — Measurement of capillary flow in the rectal microcirculation
Procedure: Urine collection (Foley catheter) — For urinalysis, biochemistry, urine microscopy, pH, and culture.
Procedure: Venous blood samplings — for: parasitological and microbiological diagnostics, complete blood count, biochemistry, red cell deformability analyzed by laser assisted rotational cell analyser (LORCA), markers of oxidative stress (peripheral intravenous catheter)
Procedure: Electrocardiogram — all patients will have an ECG performed on enrolment as a non-invasive investigation
Procedure: GlycoCheck — GlycoCheck is a clinical sublingual handheld, bedside microscope that detects erythrocytes within the small sublingual blood vessels measuring 5 to 25 micrometers in diameter. The sublingual vasculature is a validated site for measuring thickness of the endothelial glycocalyx.

SUMMARY:
Sepsis and severe malaria together contribute to an estimated 13 million deaths annually, a great burden of which is in low-income countries. Optimal fluid management is critical yet remains one of the most challenging clinical care elements as volume overload precipitates pulmonary edema and volume restriction may exacerbate acute kidney injury. These complications of sepsis and severe malaria significantly increase mortality, particularly in resource-limited settings lacking mechanical ventilation and renal replacement therapy. Point-of-care ultrasound and passive leg raise testing are two easily implementable, safe and non-invasive clinical bedside fluid assessment tools that could be applied towards developing a fluid management algorithm in low resource settings. Similarly, simple tissue perfusion measures can facilitate understanding of precise indications or contraindication to fluid and vasopressor therapy.

However, the performance of these tools has yet to be confirmed in these settings. Accurate assessment of pulmonary tolerance and fluid responsive patients could aid to tailor vasopressor and fluid therapy to the patient condition and disease phase, thus preventing or detecting iatrogenic pulmonary edema and other pulmonary complications. As there is currently limited evidence supporting fluid management recommendations for severe malaria and sepsis in low-resource settings, the potential application of these management tools could optimize supportive therapy and improve outcomes in these populations.

The main activity proposed is a prospective, observational study of patients with sepsis and severe malaria to describe the relationship between fluid therapy and vasopressor therapy against measures of tissue perfusion and pulmonary congestion in adult patients with severe malaria or severe sepsis. In addition, the study will assess the performance of simple bedside clinical tools assessing fluid responsiveness, pulmonary congestion and peripheral tissue perfusion.

The data from this observational study will facilitate the preparation of a follow-up study to test a clinical algorithm to guide individualized fluid and vasopressor administration.

DETAILED DESCRIPTION:
This will be a single center, prospective, longitudinal, observational study of patients with sepsis or severe malaria. It is planned that this initial observational study will inform a follow-up intervention study, based on the observational study findings (Lung Ultrasound and Passive Leg Raising- guided Vasopressors and Fluid Management in Patients with Sepsis and Severe Malaria). The follow-up study will propose testing of a clinical algorithm to individualize titration of vasopressors, diuretics and fluids based on the simple tools evaluated during the observational study.

The expected duration of study patient participation is 30 days. Patients will be assessed every 6 hours until fever clearance, parasite clearance (in malaria patients) and GCS normalization (score of 15) on two consecutive assessments. Thereafter, patients will be assessed daily until discharge or death with one follow-up visit at 14 days and a follow-up call at day 30. The prospective, observational recruitment phase of the study is expected to last 15 months.

Funder: Wellcome Trust of Great Britain, Grant reference number: 220211/A/20/Z

ELIGIBILITY:
Inclusion Criteria:

I. Sepsis criteria:

The sepsis criteria include the severe sepsis and septic shock categories according to 2012 Surviving Sepsis Campaign guidelines. Due to a possible delay in obtaining all the enrolment sequential organ failure assessment (SOFA) score variables necessary to fulfil the criteria for the latest 2016 sepsis definition, the 2012 Surviving Sepsis Campaign criteria and the quick SOFA tool will be used for inclusion. However, after study completion, when all admission SOFA scores will be available, all patients will be re-scored according to the Sepsis 3 definition.

Inclusion criteria for sepsis:

1. Documented or suspected infection
2. Systolic blood pressure ≤ 100 mmHg, or receiving vasopressor (epinephrine, norepinephrine, dopamine)

   PLUS one or more of the following:

   A. Respiratory rate ≥22 breaths per minute or under oxygen therapy or mechanical ventilation B. Altered mental status (Glasgow Coma Scale ≤ 14)
3. Fully informed written consent obtained, including written informed consent from a relative or parent/guardian in case of reduced consciousness and/or age < 16 years.
4. Age ≥12 years
5. Negative peripheral blood slide for any stages of malaria parasites and a negative rapid diagnostic test (RDT) for falciparum and vivax malaria.
6. Within 24 hours of hospital or ICU admission

Note: Positive blood or urine cultures not required as eligibility criteria due to limited microbiology laboratory availability.

II. Severe malaria criteria Using modified World Health Organization criteria for severe falciparum malaria, as defined previously.

* Any P. falciparum or P. vivax parasitaemia in adults, detected by asexual stages on a peripheral blood- slide or a positive RDT in combination with one or more:

  i. GCS <11 ii. Hematocrit < 20% with parasite count >100,000/mm3 iii. Jaundice with parasite count >100,000/mm3 iv. Serum creatinine >3 mg/dL (or anuria) v. Hypoglycemia with venous glucose <40 mg/dL vi. Systolic blood pressure <80 mmHg with cool extremities vii. Peripheral asexual stage parasitemia >10 % viii. Peripheral venous lactate >4 mmol/L ix. Peripheral venous bicarbonate <15 mmol/L x. Respiratory distress/pulmonary edema: radiologically confirmed, or oxygen saturation <92% on room air with a respiratory rate >30/min, often with chest indrawing and crepitations on auscultation xi. Spontaneous bleeding xii. Generalized convulsions (≥2 in 24 hours)
* Fully informed written consent obtained, including written informed consent from relative or parent/guardian in case of reduced consciousness and/or age < 16 years.
* Age ≥12 years
* Within 24 hours of antimalarial treatment

III. Uncomplicated malaria criteria (control group)

* P. falciparum slide positive (asexual stages) on peripheral blood slide or positive RDT in combination with none of the above severity criteria.
* Within 24 hours of start of antimalarial treatment
* Fully informed written consent obtained, including written informed consent from relative or parent/guardian in case of reduced consciousness and/or age < 16 years.
* Age ≥12 years

Exclusion Criteria

The participant may not enter the study if ANY of the following apply:

* Patients admitted with known malignancy or liver disease
* Recent surgery (as part of current admission)
* Trauma (resulting in current admission)
* Antimalarial treatment ≥24 hours prior to screening

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female subjects, aged ≥12 years hospitalized with malaria or sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Fluid balance volume at 24 hours | On the first 24 hours from enrollment
  Fluid balance volume in milliliters calculated daily as inputs minus outputs.
Plasma lactate levels | 72 hours
  Plasma venous lactate levels expressed in mmol/L
Vasopressor therapy | 72 hours
  Expressed as dichotomous variable, use of any vasopressor during the first 72 hours.
Global ultrasound aeration score | 72 hours
  The score ( range 0-36) is calculated over 12 lung zones where each zone is scored 0 to 3.
Fluid balance volume at 48 hours | On the first 48 hours from enrollment
  Fluid balance volume in milliliters calculated daily as inputs minus outputs.
Fluid balance volume at 72 hours | On the first 72 hours from enrollment
  Fluid balance volume in milliliters calculated daily as inputs minus outputs.

SECONDARY OUTCOMES:
Plasma creatinine levels | 48 hours
  Measured in millimoles per liter.
Positive chest X-ray for pulmonary edema (dichotomous variable) | 72 hours
  Other measures evaluating pulmonary congestion
The ratio between pulse oxymetry hemoglobin saturation and the fraction of inspired oxygen (SpO2/FiO2 ratio). | 72 hours
  Other measures evaluating pulmonary congestion
Proportion of fluid responsive patients | 72 hours
  Fluid responsiveness is defined as a positive pulse pressure passive leg raise test (change in pulse pressure >10% after leg raise manouver) or cardiac output-guided passive leg raise test (change in cardiac output >10% after leg raise manouver). The passive leg raise test is performed both a standard maneuver (bed tilting) and a modified maneuver (manual leg raise).
Prolonged capillary refill time (dichotomous variable, defined as ≥3 seconds) | 72 hours
  Other measures evaluating tissue perfusion
Skin mottling score (0-5) | 72 hours
  Other measures evaluating tissue perfusion
Cardiac index (in liters per minute per square meter of body surface area) | 72 hours
  Other measures evaluating tissue perfusion
Core-periphery temperature gradient(°C) | 72 hours
  Other measures evaluating tissue perfusion
Proportion of patients at enrolment and during admission with a low cardiac index and hypoperfusion state. | 72 hours
Proportion of patients with microvasculature obstruction or abnormalities | 24 hours
  Microvasculature obstruction and abnormalities are detected with orthogonal polarization spectral imaging (OPS); red cell deformability is studied by laser assisted rotational cell analyser (LORCA).
Proportion of patients that develop pulmonary edema and acute respiratory distress syndrome (ARDS). | 72 hours
  Pulmonary edema is defined as the presence of 2 or more positive lung zones per hemithorax on the lung ultrasound. Acute respiratory distress syndrome is defined according to the Berlin Definition criteria.
Case fatality in first 30 days. | 30 days
Acute kidney injury (AKI) | At admission, up to day 14, and renal recovery by 30 days
  Proportion of AKI as per Kidney Diseases Improving Global Outcomes definition: serum creatinine increase by ≥ 3 mg/dl within 48 hours, or serum creatinine increase by ≥ 1.5 times baseline, or urine volume <0.5 mg/kg/h for 6 hours. Outcome of AKI defined as renal recovery (time in days until creatinine returns to baseline).
Proportion of patients that develop lower extremity deep venous thrombosis. | 72 hours
  Deep venous thrombosis is defined as a positive compressive ultrasonography on femoral or popliteal veins of lower limbs.
Microbiological etiology of sepsis. | 72 hours
  Results of blood culture and organism identified in case of positive result
Number of patients with ARDS according to the Kigali Modification of the Berlin Definition of ARDS | 72 hours
Diagnostic performance measures (sensitivity, specificity, positive predictive value, negative predictive value) of the digital microscope with expert microscopy as the gold standard | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Chittagong Medical College Hospital, Chittagong, Bangladesh